CLINICAL TRIAL: NCT03156673
Title: Primary Research on Treatment of Chronic Obstructive Pulmonary Disease (COPD) by Transplantation of Autologous Bronchial Basal Cells
Brief Title: Treatment of COPD by Autologous Transplantation of Bronchial Basal Cells
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Shantou University Medical College (Other)
Collaborators: Regend Therapeutics (Industry); Tongji University (Other)
Responsible Party: Principal Investigator, Xiaohe Zheng, Chief Physician, First Affiliated Hospital of Shantou University Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017112
Record Dates: First submitted 2017-05-13; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bronchial basal cells (Experimental): Patients will receive of clinical grade bronchial basal cells (BBCs) with a dosage of 10^6 (1 million) cells/Kg/person via fiberoptic bronchoscopy after fully lavage of the localized lesions.
  Interventions: Biological: bronchial basal cells

INTERVENTIONS:
Biological: bronchial basal cells — Patients will receive of clinical grade bronchial basal cells (BBCs) with a dosage of 10^6 (1 million) cells/Kg/person via fiberoptic bronchoscopy after fully lavage of the localized lesions.

SUMMARY:
Bronchial basal cells are proved to be able to regenerate lung structures to repair the injured lung. In COPD patients, bronchus structures are injured and cannot be repaired, which may result in the failure of pulmonary function rescue clinically.In our research, autologous bronchial basal cells will be transplanted into lung of patients suffered with COPD to treat the disease. Specifically, autologous bronchial basal cells will be dissected from brushed-off samples by bronchofiberscope. Then, they will be expanded in vitro and transplanted into lung to regenerate new alveoli and bronchus structures and re-establish pulmonary system.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40 to 75;
* Diagnosed with COPD according the guideline (a. with symptoms of productive cough, sputum production or shortness of breath; b. with poor airflow as indicated by FEV1<70% predicted value and FEV1/FVC < 0.7 in pulmonary function test; c. with exclusion of other pulmonary disease by CT or blood examination);
* Clinically stable for more than 4 weeks;
* Tolerant to bronchofiberscope;
* Written informed consent signed.

Exclusion Criteria:

* Pregnant or lactating women;
* Patients positive for syphilis, HIV;
* Patients with malignant tumor;
* Patients with serious or significant pulmonary infection and need anti-infection treatment;
* Patients with serious heart disease(NYHA class Ⅲ-Ⅳ);
* Patients with a history of abusing alcohol and illicit drug;
* Patients participated in other clinical trials in the past 3 months;
* Patients assessed as inappropriate to participate in this clinical trial by investigator.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | 1-6 months
  An indicator for pulmonary function test to assess airway obstruction
Forced vital capacity (FVC) | 1-6 months
  An indicator for pulmonary function test to indicate the maximum amount of air a person can expel from the lungs after a maximum inhalation

SECONDARY OUTCOMES:
Diffusion capacity of CO (DLCO) | 1-6 months
  An indicator for pulmonary function test to show the extent to which oxygen passes from the air sacs of the lungs into the blood
The ratio of forced expiratory volume in the first one second to the forced vital capacity (FEV1/FVC) | 1-6 months
  An indicator in pulmonary function test to represent the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration to the full vital capacity
Maximum mid-expiratory flow (MMF) | 1-6 months
  An indicator in pulmonary function test to stand for maximal (mid-)expiratory flow and is the peak of expiratory flow as taken from the flow-volume curve and measured in liters per second
Maximum voluntary ventilation (MVV) | 1-6 months
  An indicator in pulmonary function test to measure the maximum amount of air that can be inhaled and exhaled within one minute
6-minute-walk test (6MWT) | 1-6 months
  An indicator to evaluate the exercise function of patients with moderate or severe pulmonary heart diseases
Modified medical research council (MMRC) chronic dyspnea scale | 1-6 months
  An indicator to evaluate the level of dyspnea
St. George's respiratory questionnaire (SGRQ) scale | 1-6 months
  A questionnaire to assess life quality affected by the respiratory problems

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No